CLINICAL TRIAL: NCT02877199
Title: Anti-E1E2 Antibodies for the Prediction of Virological Response to Triple Therapy in Treatment-experienced Hepatitis C Virus-cirrhosis Cases
Brief Title: Anti-E1E2 Antibodies (D32.10 Epitope-binding Antibodies) and HCV Triple Therapy
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0552
Record Dates: First submitted 2016-08-12; First posted 2016-08-24 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; anti-E1E2 antibodies; cirrhosis; triple therapy
MeSH Terms: conditions — Hepatitis C; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- HCV triple therapy: Cohort of HCV patients who received first-generation protease inhibitor-based triple therapy
  Interventions: Other: Triple therapy

INTERVENTIONS:
Other: Triple therapy — Cohort of patients who received triple therapy combining pegylated-interferon/ribavirin + first generation protease inhibitor boceprevir or telaprevir as part of routine clinical practice

SUMMARY:
The hypothesis was to check whether baseline anti-E1E2 antibodies were correlated with the on-treatment viral kinetics and could predict virological outcome in treatment-experienced HCV-infected cirrhotic patients receiving protease inhibitor-based triple therapy.

ELIGIBILITY:
Inclusion Criteria:

* HCV patients with compensated cirrhosis (Child-Pugh A)
* HCV genotype 1
* non-responders to a previous course of interferon (IFN)/ribavirin
* receiving boceprevir or telaprevir

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatitis C virus infected patients with cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with positive anti-E1E2 antibody level at treatment initiation | Baseline (initiation of treatment)
  Anti-E1E2 antibody levels were determined as previously described (Ndongo et al. Hepatology 2010;52:1531-42) using optical densities obtained after dilution of patients' serum samples at 1/250 and 1/500. Samples with anti-E1E2 levels above 950 (OD value× 1000) were considered positive.

SECONDARY OUTCOMES:
Kinetic of Quantification of hepatitis C viral load (HCV RNA) | baseline (initiation of treatment), at week 4, 12, 24, 36, 48 of therapy, at 12 weeks after the end of treatment.
  Viral load was assessed at baseline (initiation of treatment), and at week 4, 12, 24, 36, and 48 of therapy and 12 weeks after the end of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de la Croix Rousse, Lyon, France